CLINICAL TRIAL: NCT03365557
Title: A Clinical Study of the Setting of Laryngeal Mask Airway Intracuff Pressure Based on Airway Peak Pressure
Brief Title: Airway Peak Pressure-directed Laryngeal Mask Airway Intracuff Pressure Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Zhuan Zhang, Principal Investigator, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20171110
Record Dates: First submitted 2017-11-10; First posted 2017-12-07 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2017-12

CONDITIONS: Laryngeal Mask Airway

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intracuff pressure set by airway peak pressure (Experimental)
  Interventions: Procedure: Airway peak pressure
- Intracuff pressure set at 60 mmHg (Other)
  Interventions: Procedure: Airway peak pressure

INTERVENTIONS:
Procedure: Airway peak pressure — Air was injected into LMA cuff during expiration phase to make intracuff pressure achieve the level of airway peak pressure. If there's any leakage, increase 5 cmH2O every time till there's no air leakage from the mouth.

SUMMARY:
The investigators aimed to explore the effects of airway peak pressure (Ppeak) guidance on the least laryngeal mask airway (LMA) intracuff pressure setting during general anesthesia and the effects on postoperative complications in the throat. One hundred and twenty patients (American Society of Anesthesiologists grades I or II) scheduled for elective laparoscopic cholecystectomy under general anesthesia were enrolled in our study. The patients were divided into pressure-regulated group (group P) and control group (group C) randomly. Supreme LMA was inserted in after general anesthesia induction. Air was injected into the cuff to make the intracuff pressure (ICP) achieve 60 cmH2O. Volume-controlled ventilation was selected and Ppeak was recorded. In group P, all the gas in the LMA cuff was sucked out, and then air was injected in during expiration phase to make ICP achieve the level of Ppeak. If there's any leakage, increase 5 cmH2O every time till there's no air leakage from the mouth. After pneumoperitoneum, the cuff was inflated to make ICP achieve 60 cmH2O and Ppeak was recorded once more. Then all the gas in the LMA cuff was sucked out, and air was injected into the cuff during expiration phase to make ICP achieve the level of Ppeak as the above method till the end of operation. During pneumoperitoneum, the pressure of CO2 was set at 10 cmH2O. In group C, ICP was maintained at 60 cmH2O. Ppeak, ICP and the intracuff gas volume were recorded before and after pneumoperitoneum. ICP during inspiratory phase in the two groups was measured. Tidal volume during inspiration (VTI) and expiration (VTE) in the two groups were recorded, and the leakage rate was calculated as [(VTI-VTE)/ VTI×100%]. Throat complications of all the patients in 24 hours after surgeries were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiologists grades I or II scheduled for elective laparoscopic cholecystectomy under general anesthesia

Exclusion Criteria:

* Patients with limited head and neck activity, limited mouth opening, high abdominal pressure, inflammation of the throat and respiratory diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
The intracuff gas volume before pneumoperitoneum | Intraoperative
  The changes of intracuff gas volume before pneumoperitoneum
The intracuff gas volume after pneumoperitoneum | Intraoperative
  The changes of intracuff gas volume after pneumoperitoneum
The intracuff pressure before pneumoperitoneum | Intraoperative
  The changes of intracuff pressure before pneumoperitoneum
The intracuff pressure after pneumoperitoneum | Intraoperative
  The changes of intracuff pressure after pneumoperitoneum

SECONDARY OUTCOMES:
Throat complications | From the end of operation till 24 hs postoperative
  Throat pain, swallow discomfort and hematoma